CLINICAL TRIAL: NCT03297606
Title: Canadian Profiling and Targeted Agent Utilization Trial (CAPTUR): A Phase II Basket Trial
Brief Title: Canadian Profiling and Targeted Agent Utilization Trial (CAPTUR)
Acronym: CAPTUR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry); Bristol-Myers Squibb (Industry); Hoffmann-La Roche (Industry); Pfizer (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1; ESR-17-12831 (Other: AstraZeneca); CA209-9DL (Other: Bristol-Myers Squibb); ML39800 (Other: Hoffmann-La Roche); WI233446 (Other: Pfizer)
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma; Advanced Solid Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — olaparib; Dasatinib; Nivolumab; Ipilimumab; Axitinib; bosutinib; Crizotinib; palbociclib; Sunitinib; temsirolimus; Erlotinib Hydrochloride; Trastuzumab; pertuzumab; Vemurafenib; cobimetinib; HhAntag691; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Group 1 - Arm CLOSED, no patients recruited (Experimental): VEGFR1, VEGFR2, VEGFR3
  Interventions: Drug: Axitinib
- Group 2 - Arm CLOSED, no patients recruited (Experimental): BCR-ABL, SRC
  Interventions: Drug: Bosutinib
- Group 3 - Arm CLOSED (Experimental): ALK, ROS1, MET
  Interventions: Drug: Crizotinib
- Group 4 - Arm CLOSED, no patients recruited (Experimental): KIT, PDGFRA, PDGFRB, ABL1
  Interventions: Drug: Dasatinib
- Group 5 - Arm CLOSED (Experimental): EGFR
  Interventions: Drug: Erlotinib
- Group 6 - Arm CLOSED (Experimental): high mutation burden, POLE, POLD1
  Interventions: Drug: Nivolumab plus Ipilimumab
- Group 7 - Arm CLOSED (Experimental): BRCA1, BRCA2, mutations in HRD
  Interventions: Drug: Olaparib
- Group 8 - Arm CLOSED (Experimental): CDKN2A, CDK4, CCND1, SMARCA4
  Interventions: Drug: Palbociclib
- Group 9 Arm CLOSED (Experimental): CSF1R, PDGFRA, PDGFRB,VEGFR1, VEGFR2, VEGFR3, KIT, FLT3, RET, FGFR1, FGFR2, FGFR3, VHL
  Interventions: Drug: Sunitinib
- Group 10 Arm CLOSED (Experimental): AKT1, AKT2, AKT3, FBXW7, FLCN, mTOR, NF1, NF2, NTRK3, PIK3CA, PIK3R1, PTEN, RHEB, STK11, TSC1, TSC2
  Interventions: Drug: Temsirolimus
- Group 11 - Arm CLOSED (Experimental): ERBB2
  Interventions: Drug: Trastuzumab plus Pertuzumab
- Group 12 - Arm CLOSED (Experimental): BRAFV600
  Interventions: Drug: Vemurafenib plus Cobimetinib
- Group 13 - Arm CLOSED (Experimental): PTCH1, SMO
  Interventions: Drug: Vismodegib
- Group 14 (Experimental): ERBB2
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Olaparib — 300mg taken twice daily
  Arms: Group 7 - Arm CLOSED
Drug: Dasatinib — 100mg administered orally once daily
  Arms: Group 4 - Arm CLOSED, no patients recruited
Drug: Nivolumab plus Ipilimumab — * Combination Phase - 3mg/kg nivolumab administered as an intravenous infusion over 30 minutes every 3 weeks for the first 4 doses in combination with ipilmumab 1mg/kg administered intravenously over 30 minutes, followed by the single-agent phase.
  * Single-Agent Phase - 480mg nivolumab administered as an intravenous infusion over 30 minutes every 4 weeks.
  Arms: Group 6 - Arm CLOSED
Drug: Axitinib — 5mg orally twice daily
  Arms: Group 1 - Arm CLOSED, no patients recruited
Drug: Bosutinib — 500mg orally once daily
  Arms: Group 2 - Arm CLOSED, no patients recruited
Drug: Crizotinib — 250mg orally twice daily
  Arms: Group 3 - Arm CLOSED
Drug: Palbociclib — 125mg orally once daily for 21 consecutive days followed by 7 days off treatment to comprise a complete cycle of 28 days
  Arms: Group 8 - Arm CLOSED
Drug: Sunitinib — 50mg orally once daily on a schedule of 4 weeks on treatment followed by 2 weeks off
  Arms: Group 9 Arm CLOSED
Drug: Temsirolimus — 25mg infused over a 30-60 minute period once a week
  Arms: Group 10 Arm CLOSED
Drug: Erlotinib — 150mg orally, once daily
  Arms: Group 5 - Arm CLOSED
Drug: Trastuzumab plus Pertuzumab — Trastuzumab = 3-weekly dose schedule. The recommended initial loading dose is 8mg/kg administered as a 90-minute infusion followed by 3-weekly maintenance dose of 6mg/kg administered as 90-minute infusion.
  Pertuzumab = 840mg administered as a 60-minute intravenous infusion, followed every 3 weeks thereafter by a dose of 420mg administered over a period of 30-60 minutes.
  Arms: Group 11 - Arm CLOSED
Drug: Vemurafenib plus Cobimetinib — Vemurafenib = 960 mg orally every 12 hours.
  Cobimetinib = 60 mg orally once daily for 21 days, followed by 7 days of rest
  Arms: Group 12 - Arm CLOSED
Drug: Vismodegib — 150mg taken orally, once daily
  Arms: Group 13 - Arm CLOSED
Drug: Tucatinib — 300mg taken orally, twice daily
  Arms: Group 14

SUMMARY:
Cancer drugs which target the effects of abnormal gene changes are called 'targeted therapies'. This study, called PM.1 or CAPTUR, will include some targeted therapies that are currently available. The purpose of this study is to find out what are the effects on a patient and their cancer when they are given a targeted therapy drug that is specific to an abnormal gene change in their cancer.

DETAILED DESCRIPTION:
Recent advances in laboratory technology have enabled the identification of changes in the genetic makeup of tumors that might be responsible for their malignant behavior such as uncontrolled growth and spread. Some of these changes can be 'druggable', i.e. there may be cancer medicines that can specifically act on the tumour's genetic abnormality. Several cancer centers and programs have initiated this type of molecular profiling across Canada, with the goal to identify 'druggable' changes in tumors to find matching therapy for patients. These include initiatives in British Columbia, Ontario and Quebec. The CAnadian Profiling and Targeted agent Utilization tRial (CAPTUR) will test the activity of a list of commercially available targeted agents in patients who have undergone tumor profiling and have 'druggable' changes identified in their cancers.

ELIGIBILITY:
Inclusion Criteria: (screening step - non-drug specific)

* Adult (≥ 18 yrs) patient with a histologically-proven incurable metastatic solid tumour (excluding primary brain tumours), multiple myeloma or B cell non-Hodgkin lymphoma (excluding CLL, SLL and HCL), for whom there is no standard treatment known to prolong life, or who has refused such treatment.
* ECOG performance status 0-2.
* Patients must have normal organ function as follows:

  * Absolute neutrophil count: ≥ 1.5 x 10^9/L for solid tumours; ≥ 1.0 x 10^9/L for neurologic malignancies
  * Platelets ≥ 75 x 10^9/L (or ≥ 50 x 10^9/L if bone marrow involvement by myeloma or lymphoma).
  * Total bilirubin ≤ 1.5 x UNL.
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal value unless liver metastases are present in which case they must be < 5 x ULN;
  * Serum creatinine ≤ 1.5 x UNL or calculated or measured creatinine clearance ≥ 50mg/min/1.73µ^2
* Patients must have measurable disease
* Results must be available from tumour genomic or protein expression testing (if used to identify genetic variants), from one of the initiatives / groups listed in protocol Appendix VII. The test may have been performed on the primary tumour or a metastatic deposit (including bone marrow), or blood, in a diagnostic or research laboratory and must reveal a potentially actionable variant.
* Patient consent (Main Study Consent for the screening step) must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to the screening step to document their willingness to participate
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre or a CCTG IND site. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria: (screening step - non-drug specific)

* Patients with prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Patients with ongoing toxicity ≥ CTCAE grade 2, other than peripheral neuropathy or asymptomatic, corrected biochemical toxicities (e.g. hypothyroidism corrected by thyroid replacement), related to prior anti-tumour treatment. Patients with ongoing peripheral neuropathy of ≥ CTCAE grade 3 will be excluded.
* Patients concurrently receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g. megestrol acetate, bisphosphonates) or ongoing castration-intent therapy for prostate cancer. These medications must have been started ≥ one month prior to enrollment on this study. Patients may be on warfarin, low molecular weight heparin or direct factor Xa inhibitors, unless such therapies are prohibited by drug-specific ineligibility criteria.
* Patients with known active progressive brain metastases. Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within one month prior to screening. All patients with previously treated brain metastases must be stable (clinically and radiologically) for at least one month after completion of treatment and either off steroid treatment or only taking physiological doses of steroids prior to the screening step.
* Patients with clinically significant pre-existing cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure.
* Patients with known left ventricular ejection fraction (LVEF) < 40%.
* Patients with stroke (including TIA) or acute myocardial infarction within three months prior to the screening step.
* Patients with acute gastrointestinal bleeding within one month prior to the screening step.
* Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations.
* Lactating and nursing women
* Patients who do not meet drug-specific eligibility requirements for the drug selected by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate defined as the number of patients with complete response or partial response | 4 years
  over the total number of patients in a given cohort.

SECONDARY OUTCOMES:
Number and severity of adverse events grade >3, or of lesser grade resulting in discontinuation, delay or reduction in dose of study drug | 4 years
  measured by CTCAE
Progression-free survival by disease-appropriate objective criteria | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Study Chair — Univ. Health Network-OCI/Princess Margaret Hospital, Toronto, ON Canada; Daniel J Renouf, Study Chair — BCCA - Vancouver Cancer Centre, Vancouver BC, Canada
Locations (10):
- Canada (10):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy
URL: https://www.ctg.queensu.ca/public/policies